CLINICAL TRIAL: NCT05133661
Title: Feasibility and Acceptability of Implementing Integrated HPV Testing and Treatment of Pre-cancerous Cervical Cancer Lesions in Burkina Faso, Côte d'Ivoire, Guatemala, and the Philippines
Brief Title: SUCCESS - Feasibility of HPV Testing and Treatment of Pre-cancerous Cervical Cancer Lesions (HPV Study)
Acronym: HPV
Status: Active, not recruiting | Type: Observational
Sponsor: Jhpiego (Other)
Collaborators: UNITAID (Other); Expertise France (Other); World Health Organization (Other)
Responsible Party: Principal Investigator, Mark Kabue, Sr. Monitoring Evaluation and Research Advisor, Jhpiego
Other Study IDs: ERC0003618; IRB13630 (Other: Johns Hopkins Bloomberg School of Public Health IRB)
Record Dates: First submitted 2021-11-13; First posted 2021-11-24 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer
Keywords: HPV Screening; Precancerous lesions; Thermal ablation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HPV positive women: Women aged 25-49 years seeking offered HPV testing (either self-collection or clinician collection of samples) and treatment of precancerous lesions as part of service package in study facilities will be enrolled in the study and interviewed at different time points.
  A subset of the women screened will be selected for in-depth interview to gather data on: ease of use of self-collection kits for cervical cancer screening, receipt of the test results, and treatment for precancer. Another subset of women will be selected after HPV screening to participate in client exit interview.
  Interventions: Diagnostic Test: HPV testing

INTERVENTIONS:
Diagnostic Test: HPV testing — Interviews will be conducted among women from the general population and HIV+ women after screening for HPV. A small subset of participants will be interviewed after receiving treatment for precancer. HPV test results and outcome of the precancer treatment if indicated will be documented.
  Other Names: Thermal ablation of precancerous lesion

SUMMARY:
The goal is to assess the feasibility and acceptability of integrating into existing health systems, provision of HPV screening and treatment of pre-cancerous cervical cancer lesions with ablative treatments in Burkina Faso, Côte d'Ivoire, Guatemala, and the Philippines. Study findings will inform implementation of cervical cancer prevention and treatment services as part of a global effort to eliminate cervical cancer, with particular relevance for low-and-middle income countries. This will inform country strategy and guidelines on offering integrated cervical cancer prevention and treatment services in a manner that is culturally sensitive, client oriented, and system appropriate.

DETAILED DESCRIPTION:
Research question:

1. How feasible is it to implement integrated HPV testing (including self-collection of samples) and ablative treatment of lesions precancerous cervical cancer lesions among HPV+ women aged 30-49 years (general population) and 25-49 years (WLHIV), leveraging on the existing health systems in the four study countries?
2. What is the acceptability of HPV screening through self-collection or clinician collection of sample, and ablative treatment of precancerous lesions among women accessing cervical cancer services in the study sites?
3. What is the cost of implementing integrated cervical cancer screening and precancer treatment services (Supply: counselling, HPV testing, treatment, training health care providers, etc.), and user-related costs (travel, out of pocket expenses opportunity costs, etc.) in the SUCCESS project supported sites?
4. Which factors influence the successful implementation of integrated HPV screening and treatment services (e.g. perceptions, experience of care, religious beliefs, culture, individual characteristics, availability of services, cost, etc.)?

Methodology:

We will utilize a hybrid effectiveness implementation Type III study design, using mixed methods approach. In Phase I, 2,227 women are enrolled in health facilities in each of the four countries (disaggregated by general population and WLHIV) and follow those who are HPV positive to determine the completion of screen-to-treat within three months. In Phase II focusing on community self-sampling, 8,694 are enrolled in Burkina Faso, Guatemala and the Philippines.

Quantitative and qualitative data will be collected from clients, service providers, key stakeholders, and secondary analysis of service delivery including laboratory data will be analyzed to assess acceptability and feasibility of implementing integrated cervical cancer screening and treatment services.

ELIGIBILITY:
Inclusion Criteria:

* Women: Participants will be women residing in the study area, seeking services at SUCCESS project-supported health facilities, and meet the eligibility criteria to be enrolled in one of the components of the study (i.e, prospective component, client exit interviews and/or in-depth interviews).
* Service providers: Health care personnel working in the project facilities at the time of the study providing services related to cervical cancer screening and treatment. Facility in-charges and laboratory personnel are included in this category.
* Key informants: Health program managers, and community mobilizers at either local or national level in Burkina Faso, Cote d'Ivoire, Guatemala, and Philippines.
* Men: Male members of the community (married or cohabiting with female partners) to gather their perspectives on the implementation of the cervical cancer prevention and treatment activities.

Exclusion Criteria:

* Pregnant women
* Individuals unwilling to participate or unable to provide informed consent

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women screened for HPV
Study Population: * Women: Participants will be drawn from women seeking care at the SUCCESS project supported sites. For the general population, women aged 30-49 years will be enrolled while for HIV+ women, those aged 25-49 years will be enrolled. Women who do not know their HIV status at enrolment will have an opportunity to be tested.
  * Key informants will be identified from among the stakeholder holding positions that allows them to provide information that is relevant to the assessment of acceptability, feasibility, and costs related to implementation of cervical cancer prevention and treatment services in the four countries. from seeking care in health facilities in the four countries.
Sampling Method: Non-Probability Sample
Enrollment: 17602 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of HPV positive women who complete screen to treatment within 3 months | Three months
  Proportion of HPV positive women who undergo treatment for precancerous cervical lesions within three months of screening

SECONDARY OUTCOMES:
Acceptability - Percentage of women screened for HPV who report positive experience of care | 18 months
  Assess the adoption, satisfaction, and uptake of the cervical cancer services by the users and the providers
Feasibility - Turnaround time from screening to treatment | 18 months
  Assess the adoption and practicability of providing the cervical cancer services through the mechanisms that exist in of each of the four countries
Unit cost of providing HPV screening and treatment of precancerous cervical cancer lesion | 18 months
  The cost of providing the services and the user costs

CONTACTS AND LOCATIONS:
Locations (4):
- CMA de Do, Ouagadougou, Burkina Faso
- FSU Koko, Bouaké, Côte d’Ivoire
- Quetzaltenango, Quetzaltenango, Guatemala
- Metro-Manila, Quezon City, Philippines, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kabue M, Gauvreau CL, Daceney N, Bertram MM, Shissler T, Reis V, Dodo M, Garces A, Llave C, Dao B, Mohan D, Huang L. Understanding integrated HPV testing and treatment of pre-cancerous cervical cancer in Burkina Faso, Cote d'Ivoire, Guatemala and Philippines: study protocol. Reprod Health. 2023 Nov 13;20(1):167. doi: 10.1186/s12978-023-01696-8. PMID 37957689